CLINICAL TRIAL: NCT00551902
Title: Effect of an Anterior Chamber Infusion System on Trabeculectomy Outcomes
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Efficacy study indicated that further study is not warranted
Sponsor: Queen's University (Other)
Collaborators: Glaucoma Research & Education Group (Other)
Responsible Party: Principal Investigator, Dr. Robert Campbell, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC-2
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Glaucoma
Keywords: Glaucoma; trabeculectomy; anterior chamber maintainer; anterior chamber infusion
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Trabeculectomy with anterior chamber infusion system
  Interventions: Procedure: Trabeculectomy with anterior chamber infusion system
- 2 (Active Comparator): Trabeculectomy without anterior chamber infusion system
  Interventions: Procedure: Trabeculectomy without anterior chamber infusion system

INTERVENTIONS:
Procedure: Trabeculectomy with anterior chamber infusion system — Trabeculectomy with anterior chamber infusion system
  Arms: 1
Procedure: Trabeculectomy without anterior chamber infusion system — Standard trabeculectomy surgery
  Arms: 2

SUMMARY:
In the treatment of glaucoma, trabeculectomy surgery provides a drainage system for the eye and allows for the lowering of the pressure inside the eye. The flow through the surgically created fistula determines the intraocular pressure. Titrating suture tightness is important to achieving the desired post-operative intraocular pressure. This process is not straightforward and intraocular pressures are often too high or too low post-operatively.

DETAILED DESCRIPTION:
The use of an anterior chamber infusion system to deliver fluid into the eye during trabeculectomy surgery may be of benefit in this process and may have other benefits as well which may result in better outcomes.

Thus, the hypothesis of this study is that the use of an anterior chamber infusion system improves success of trabeculectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* One of the following diagnoses:

  * primary open angle glaucoma
  * chronic angle closure glaucoma
  * pseudo exfoliation glaucoma
  * pigment dispersion glaucoma

Exclusion Criteria:

* unable to provide consent or return for follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
surgical success: intraocular pressure lowered by 30% and functional filtering bleb | 2 weeks, 1 month, 3 months, 6 months and 1 year post surgery

SECONDARY OUTCOMES:
Need for laser suture lysis | any point post operatively
complications: aqueous misdirection, suprachoroidal hemorrhage, anterior chamber shallowing | any time post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Campbell, MD, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Hotel Dieu Hospital, Queen's University, Kingston, Ontario
  - Toronto Western Hospital, University of Toronto, Toronto, Ontario